CLINICAL TRIAL: NCT01845064
Title: A Double-Blinded, Placebo-Controlled, Single-Dose and Multiple-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Proof of Concept of DM199 in Healthy Subjects and Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety and Effectiveness of DM199 in Healthy Subjects and Type 2 Diabetes Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DiaMedica Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMA-Clin-199-2013-001; 2013-000225-30 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-05-03 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Type 2
Keywords: type 2 diabetes; diabetes mellitus; type 2 diabetes mellitus; HbA1c; blood glucose; glucose control; DiaMedica; DM-199; DM199; recombinant human tissue kallikrein-1; tissue kallikrein-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — DM199

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Part A - SAD in healthy subjects (Experimental): A randomized, double-blinded, placebo-controlled, single ascending dose (SAD) study in healthy male and/or female subjects. Subjects will receive DM199 subcutaneously (sc).
  Interventions: Drug: DM199
- Part B - SAD in type 2 diabetic patients (Experimental): A randomized, partially double-blinded, placebo-controlled, sequential SAD study in male and/or female type 2 diabetes mellitus patients. Subjects will receive DM199 subcutaneously (sc).
  Interventions: Drug: DM199
- Part C - MAD in healthy subjects (Experimental): A randomized, double-blinded, placebo-controlled, 14-day multiple ascending dose (MAD) study in healthy male and/or female subjects each. Subjects will receive sequential doses of DM199 sc for 14 days.
  Interventions: Drug: DM199
- Part D - POC in type 2 diabetes patients (Experimental): A randomized, double-blinded, placebo-controlled, 28-day multiple-dose proof of concept (POC) study in male and/or female type 2 diabetes mellitus patients. Subjects will receive doses of DM199 sc for 28 days.
  Interventions: Drug: DM199
- Part A - Healthy subjects SAD placebo (Placebo Comparator): A randomized, double-blinded, placebo-controlled, single ascending dose (SAD) study in healthy male and/or female subjects. Subjects will receive placebo subcutaneously (sc).
  Interventions: Drug: Placebo
- Part B - Type 2 diabetic patients SAD placebo (Placebo Comparator): A randomized, partially double-blinded, placebo-controlled, sequential SAD study in male and/or female type 2 diabetes mellitus patients. Subjects will receive placebo subcutaneously (sc).
  Interventions: Drug: Placebo
- Part C - Healthy subjects MAD placebo (Placebo Comparator): A randomized, double-blinded, placebo-controlled, 14-day multiple ascending dose (MAD) study in healthy male and/or female subjects each. Subjects will receive placebo sc for 14 days.
  Interventions: Drug: Placebo
- Part D - Type 2 diabetic patients POC placebo (Placebo Comparator): A randomized, double-blinded, placebo-controlled, 28-day multiple-dose proof of concept (POC) study in male and/or female type 2 diabetes mellitus patients. Subjects will receive placebo sc for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DM199
  Other Names: recombinant human tissue kallikrein-1; tissue kallikrein-1
  Arms: Part A - SAD in healthy subjects; Part B - SAD in type 2 diabetic patients; Part C - MAD in healthy subjects; Part D - POC in type 2 diabetes patients
Drug: Placebo
  Arms: Part A - Healthy subjects SAD placebo; Part B - Type 2 diabetic patients SAD placebo; Part C - Healthy subjects MAD placebo; Part D - Type 2 diabetic patients POC placebo

SUMMARY:
DM199 (recombinant human tissue kallikrein-1) is a new investigational compound that may eventually be used for the treatment of Diabetes Mellitus Type 2. This is the first time that this compound is being given to humans.

The purpose of the study is to investigate to what extent DM199 is safe and tolerated. Further, it will be investigated how quickly and to what extent DM99 is absorbed and eliminated from the body (this is called pharmacokinetics). In addition, the effect of the compound on the body will be investigated (this is called pharmacodynamics).

This study is not intended to improve anyone's health, but is necessary for the further development of DM199.

The study consists of 4 parts. Each part (A, B, C and D) will consist of one or several periods. The research will be conducted in healthy male and female volunteers (Part A and C) and in male and female type 2 diabetes mellitus patients (Part B and D).

DETAILED DESCRIPTION:
DM199 (recombinant human tissue kallikrein-1) is being developed as a new biological treatment for type 2 diabetes mellitus. This is a first-in-human study for DM199 and is a 4-part, single center study in healthy subjects and type 2 diabetes mellitus patients.

Part A will be a randomized, double-blinded, placebo-controlled, single ascending dose (SAD) study in healthy male and/or female subjects. Subjects will receive DM199 or placebo subcutaneously (sc).

Part B will be a randomized, partially double-blinded, placebo-controlled, sequential SAD study in male and/or female type 2 diabetes mellitus patients.

Part C will be a randomized, double-blinded, placebo-controlled, 14-day multiple ascending dose (MAD) study in healthy male and/or female subjects each. Subjects will receive sequential doses of DM-199 or placebo sc for 14 days.

Part D will be a randomized, double-blinded, placebo-controlled, 28-day multiple-dose proof of concept (POC) study in male and/or female type 2 diabetes mellitus patients. Subjects will receive parallel doses of DM199 or placebo sc for 28 days.

The primary objective is to evaluate the safety and tolerability of single and multiple subcutaneous doses of DM199 in healthy subjects and type 2 diabetes mellitus patients. Another objective is to determine the plasma pharmacokinetic profile of DM199 after administration of single and multiple doses of DM199 in healthy subjects and type 2 diabetes mellitus patients.

Secondary objectives include determining the effect of DM199 on glucose homeostasis (via fasting glucose and HbA1c levels), standardized meal tolerance test, C-peptide, fructosamine, GLP-1 (active and total), glucagon, adiponectin and lipids measurements, and homeostatic model assessment of insulin resistance/beta cell function (HOMA) determination in type 2 diabetes mellitus patients; assessing the formation of antibodies to DM199 after administration of multiple doses of DM199 in healthy subjects and type 2 diabetes mellitus patients; and determining changes in immune cell populations by fluorescence-activated cell sorting analysis following multiple doses of DM199 in healthy subjects and type 2 diabetes mellitus patients

ELIGIBILITY:
Inclusion Criteria:

1. Status : Parts A and C: healthy subjects

   * Parts B and D: type 2 diabetes mellitus patients :
2. Body Mass Index : Parts A and C: 18.0 - 30.0 kg/m2

   * Parts B and D: 25.0 - 35.0 kg/m2
3. HbA1c : Parts B and D: at screening between 6.5% and 9.0%, inclusive for patients using one oral anti-diabetic medication, and between 6.0% and 8.5%, inclusive for patients using two or more oral anti-diabetic medications
4. Fasting blood glucose : Parts B and D: within 7.5-13.5 mmol/L, inclusive at entry into the clinical research center (Day -1 for Part B or Day -2 for Part D)
5. Women of childbearing potential agree to use an appropriate contraceptive method (hormonal, IUD, or diaphragm) until 90 days after the follow-up visit. For males: willingness to use adequate contraception from entry in the clinical research center until 90 days after the follow-up visit
6. Medical history without clinically significant abnormalities
7. Parts B and D: Taking a stable dose of one or more oral anti-diabetic medications, such as metformin, sulphonylurea or any other orally administered glucose lowering medication (except for thiazolidinediones) for at least 3 months prior to screening. Receiving no other chronic medications, including dietary supplements, that alter blood glucose control.
8. Parts A and C: Resting supine blood pressure of 140/90 mmHg or lower and higher than 90/50mmHg at screening, and showing no clinically relevant deviations as judged by the Principal Investigator
9. Parts B and D: Resting supine blood pressure of 160/100 mmHg or lower and higher than 90/50mmHg at screening, and showing no clinically relevant deviations as judged by the Principal Investigator

Exclusion Criteria:

1. Evidence of clinically relevant pathology
2. Pregnancy or lactation
3. For healthy volunteers: use of concomitant medication, except for acetaminophen (paracetamol), which is allowed up to 3 days before entry into the clinical research center (after that time the use of a limited amount of acetaminophen is permitted after consultation with the Principal Investigator). Multivitamins and vitamin C are allowed up to 7 days before entry into the clinical research center. All other medication (including over the counter medication, health supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to entry into the clinical research center.
4. Participation in a drug study within 60 days prior to drug administration. Participation in more than 3 other drug studies (for men) / more than 2 other drug studies (for women) in the 10 months preceding the start of this study)
5. Positive drug screen (opiates, methadone, cocaine, amphetamines, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants and alcohol)
6. Intake of more than 24 units of alcohol per week (one unit of alcohol equals approximately 250 mL of beer, 100 mL of wine or 35 mL of spirits)
7. Positive screen on HBsAg, anti-HCV or anti-HIV 1/2
8. Illness within 7 days prior to (the first) drug administration
9. Serum creatinine > upper limit of the normal (ULN) range

   Additional Exclusion Criteria Specific to Type 2 Diabetes Mellitus Patients (Part B and Part D)
10. The use of insulin and thiazolidinediones for type 2 diabetes mellitus 3 months prior to screening is not allowed.
11. The use of angiotensin converting enzyme (ACE) inhibitors 1 month prior to screening is not allowed.
12. History of diabetic ketoacidosis or hyperosmolar coma
13. Advanced diabetic complications, including neuropathy, nephropathy, retinopathy or other symptoms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and multiple subcutaneous doses of DM199 | Up to 13 days after final dose
  Number of participants with adverse events in the single and multiple ascending dose studies.
Determine the pharmacokinetic of DM199 after single and multiple doses | Up to 3 days after final dose
  Determine the plasma pharmacokinetic profile of DM199 after administration of single and multiple doses of DM199 in healthy subjects and type 2 diabetes mellitus patients. Measure plasma DM199 levels in individual participants.

SECONDARY OUTCOMES:
Determine the effect of DM199 on glucose homeostasis in healthy volunteers and type 2 diabetes mellitus patients | Part C, Day -1 and 14; Part D, Days -1, 14 and 28
  Determine the effect of DM199 on glucose homeostasis (via fasting glucose and HbA1c levels), standardized meal tolerance test, C-peptide, fructosamine, GLP-1 (active and total), glucagon, adiponectin and lipids measurements, and homeostatic model assessment of insulin resistance/beta cell function (HOMA) determination in type 2 diabetes mellitus patients
Assess formation of ADA to DM199 | Part C, Day -1 and 42; Part D, Day -1 and 35
  Assess the formation of antibodies to DM199 after administration of multiple doses of DM199 in healthy subjects and type 2 diabetes mellitus patients
Determine changes in immune cell populations by FACS analysis. | Part C, Day -1 and 15; Part D, Day -1 and 29
  Determine changes in immune cell populations by fluorescence-activated cell sorting analysis following multiple doses of DM199 in healthy subjects and type 2 diabetes mellitus patients

CONTACTS AND LOCATIONS:
Overall Officials: Salah Hadi, MD, MSc, Principal Investigator — PRA
Locations (1):
- PRA, Zuidlaren, Netherlands